CLINICAL TRIAL: NCT02282449
Title: Assessment of a Power Injectable vs. a Non-Power Injectable, Upper Arm, Totally Implanted Venous Access Devices for Chemotherapy
Brief Title: Power Injectable Versus a Non-Power Injectable, Upper Arm, TIVAD for Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Brent Burbridge, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-42
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malignancy
Keywords: Venous access device; Port catheters; Chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Power Injectable Port (Experimental): The subjects randomized to this group will receive the newer, power injectable port.
  Interventions: Device: Power Injectable Port (AngioDynamics Smart Port CT Mini)
- Non-Power Injectable Port (Active Comparator): The subjects randomized to this group will receive the older, non-power injectable port.
  Interventions: Device: Non-Power Injectable Port (Cook Vital Mini Port)

INTERVENTIONS:
Device: Power Injectable Port (AngioDynamics Smart Port CT Mini) — The subjects will all receive power injectable port.
  Arms: Power Injectable Port
Device: Non-Power Injectable Port (Cook Vital Mini Port) — The subjects will all receive non-power injectable port.
  Arms: Non-Power Injectable Port

SUMMARY:
Patients with cancer often require intravenous chemotherapy for long periods of time.

Ensuring that these patients have safe and reliable access to the veins for chemotherapy is challenging, and sometimes a medical device is required to administer the chemotherapy into the veins.

A totally implanted venous access device, or port, is implanted under the skin of the arm and is attached to a small plastic catheter that enters into the veins. This device can be punctured with a needle when needed for treatment or testing.

Some types of these vein ports can rapidly inject fluids (power injection), and can be used for follow-up imaging studies, such as computed tomography, that are required to follow cancer treatment effectiveness. There are no publications of randomized patients discussing the impact of power injection upon TIVAD complications and device longevity for arm implantation. The investigators propose to compare the effectiveness of power injectable against non-power injectable ports to determine if they have different clinical performance and complications. Our results will impact the care provided to cancer patients.

DETAILED DESCRIPTION:
Hypothesis:

The null hypothesis envisions both devices performing similarly in regards to chemotherapy and complications. However, the power injectable population will experience the high flow, large volume injections, may experience complications of injection extravasation and port damage due to the more vigorous injection parameters.

Trial Objectives:

1. To prospectively assess the functionality and complications of a power injectable vs. a non-power injectable TIVAD in a cohort of breast cancer patients requiring intravenous chemotherapy. The TIVAD will be randomly assigned to each patient.
2. Assess quality of life for subjects who have the two different TIVADs.
3. Facilitate device selection for future cancer patients requiring chemotherapy.

We will perform a randomized, prospective clinical trial of patients with cancer to compare a non-power injectable port, Cook Vital Mini Port (Cook Canada, Mississauga, ON), with a power injectable port, the AngioDynamics Smart Port CT Mini (AngioDynamics Inc., Manchester, GA, USA).

Adverse events, such as arm swelling, skin rash, and incision dehiscence, etc., will be tracked via an online reporting system, a patient registry, and by follow-up strategies related to imaging and clinical assessments at regular time intervals.

Patient Follow-up:

From the Insertion date, a 7 day post insertion telephone interview will be performed. Subsequently the following will be obtained at 3 months and 12 months post port insertion.

Clinical examination Venous Doppler US (arm/neck) Chest and arm X-ray QLQC30 questionnaire QLAVD-PA questionnaire Adverse Event Record

Details of Follow-up:

Clinical Examination:

Visual inspection of the arm, port implantation site, neck, and anterior chest.

1. Distended arm, neck or chest veins - Y/N - details
2. Swollen or edematous arm, neck, chest - Y/N - details
3. Skin rash - Y/N - details
4. Signs of arm infection - redness, swelling, purulent discharge - Y/N - details
5. Abnormal incision site of port insertion - Y/N - details

Venous Doppler Ultrasound (arm/neck):

Ultrasound will assess for vein thrombosis or narrowing.

Chest and arm x-rays:

Standard x-rays to include the arm from at least the elbow to axilla, full chest x-ray.

QLCC30 and QLAVD-PA:

Quality of Life surveys.

Adverse Events:

7 days, 3 months, 12 months, up to 24 months if possible - The patient will be contacted by telephone to determine if they have experienced any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients breast cancer requiring intravenous chemotherapy, referred from our local Cancer Agency for arm TIVAD, will be included.

Exclusion Criteria:

* • Those under the age of 16 years;

  * Those with uncorrectable blood clotting disorder;
  * Pregnant women, as they will not be candidates for chemotherapy;
  * Any person with an active infection or immunocompromised state;
  * Those on oral or intravenous antibiotics on the day of TIVAD implantation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Device Failure (Failure secondary to occlusion, leakage, catheter fracture, wound dehiscence) | 2 years after insertion
  Failure secondary to occlusion, leakage, catheter fracture, wound dehiscence

SECONDARY OUTCOMES:
Venous Thrombosis | 2 years after implantation
  Ipsilateral US of veins of arm and neck to detect venous thrombosis
Quality of Life Related to Port | 2 years after implantation
  Surveys of quality of life will be performed for each device
Infection | 2 years after implantation
  Detect implantation site or systemic infection related to the port.

CONTACTS AND LOCATIONS:
Overall Officials: Brent E Burbridge, MD, FRCPC, Principal Investigator — Medical Imaging, 103 Hospital Drive, Royal University Hospital, Saskatoon, SK, Canada S7N 0W8
Locations (1):
- Medical Imaging, Royal University Hospital, 103 Hospital Drive, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Goossens GA, Stas M, Jerome M, Moons P. Systematic review: malfunction of totally implantable venous access devices in cancer patients. Support Care Cancer. 2011 Jul;19(7):883-98. doi: 10.1007/s00520-011-1171-3. Epub 2011 May 10. PMID 21556721
- [Background] Marcy PY, Chamorey E, Amoretti N, Benezery K, Bensadoun RJ, Bozec A, Poissonnet G, Dassonville O, Rame M, Italiano A, Peyrade F, Brenac F, Gallard JC. A comparison between distal and proximal port device insertion in head and neck cancer. Eur J Surg Oncol. 2008 Nov;34(11):1262-9. doi: 10.1016/j.ejso.2007.09.011. Epub 2007 Nov 5. PMID 17981432
- [Background] Goltz JP, Machann W, Noack C, Hahn D, Kickuth R. Feasibility of power contrast injections and bolus triggering during CT scans in oncologic patients with totally implantable venous access ports of the forearm. Acta Radiol. 2011 Feb 1;52(1):41-7. doi: 10.1258/ar.2010.100238. PMID 21498324